CLINICAL TRIAL: NCT06318455
Title: İstanbul University-Cerrahpaşa
Brief Title: The Effect of Breathing Exercise on Sleep and Stress Levels in Women With Breast Cancer Receiving Chemotherapy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Gürcan Solmaz, Associate Professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: İstanbul University-Cerrahpaşa
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Women Receiving Chemotherapy; Poor Quality Sleep; Breast Cancer Stage II
Keywords: chemotherapy, sleep quality, breathing exercise
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises; Respiration; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breathing exercise group (Experimental): breathing exercise group: make breathing exercise for 12 weeks
  Interventions: Other: Breathing exercise
- control group (No Intervention): control group: continue standart treartment

INTERVENTIONS:
Other: Breathing exercise — For 12 weeks they will do kumbaka breathing exercise for 5 minutes twice a day in the morning and evening
  Other Names: breathing and control group
  Arms: breathing exercise group

SUMMARY:
Women receiving chemotherapy have poor sleep quality and high stress levels. With a method such as breathing exercise, which can be applied at any time without side effects, positive improvements in women's sleep and stress levels can be recorded.

DETAILED DESCRIPTION:
Women receiving chemotherapy have poor sleep quality and high stress levels. With a method such as breathing exercise, which can be applied at any time without side effects, positive improvements in women's sleep and stress levels can be recorded.

ELIGIBILITY:
Inclusion Criteria:

* women receiving chemotherapy women with poor sleep quality 18 years of age and above women with high stress levels

Exclusion Criteria:

* who do not want to participate

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the study will be conducted in women with breast cancer
Enrollment: 65 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
anxiety state scale | 12 weeks
  anxiety state scale point min:0 max:63)

CONTACTS AND LOCATIONS:
Overall Officials: Gürcan Solmaz, PhD, Study Chair — İstanbulUniversity-Cerrahpaşa; Gürcan Solmaz, PhD, Study Chair — İstanbul University-Cerrahpaşa
Locations (1):
- University of İstanbul-cerrahpaşa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No